CLINICAL TRIAL: NCT01578876
Title: To Prove up the Effect of CSWT in Vivo and to Evaluate the Feasibility and Efficiency of CSWT for Treatment of CAD and to Establish the Inclusion and Exclusion Criteria and Summarize the Methodological Outlines of CSWT in China.
Brief Title: Extracorporeal Cardiac Shock Wave Therapy (CSWT) for Treatment of Coronary Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Guo Tao, Director of Cardiovascular Center, Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSWT IN CHINA
Record Dates: First submitted 2012-02-19; First posted 2012-04-17 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; angina pectoris; myocardial ischemia; cardiac shock wave therapy
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CSWT for 3 month (Experimental): A group
  Interventions: Device: cardiac shock wave therapy(CSWT)
- CSWT for 1 month (Experimental): B group
  Interventions: Device: cardiac shock wave therapy(CSWT)
- Control group (No Intervention): C group

INTERVENTIONS:
Device: cardiac shock wave therapy(CSWT) — CSWT was performed with the MODULITH SLC SW therapy device (Storz Medical, Switzerland).Shock waves were triggered by the R-wave of the ECG when the instrument was activated. The shock wave energy was increased from an initial low level up 0.09 mJ/mm2 if the patient experienced no discomfort such as chest pain. Point-to-point combination treatment for the ischemic areas with 200 pulses delivered to each point was given.
  Other Names: SW
  Arms: CSWT for 1 month; CSWT for 3 month

SUMMARY:
The purpose of this study is to determine the effectiveness of cardiac shock wave therapy (CSWT) for the treatment of severe coronary artery disease (CAD) in a Chinese cohort.

DETAILED DESCRIPTION:
This study was approved by the Institutional Review Board and Ethics Committee of 1st Hospital of Kunming Medical University, and all study subjects signed informed consent for participation in the study and all treatments performed. Subjects were patients who were hospitalized at Department of Cardiology of our hospital from December 2008 to December 2009.

Patients were eligible to be included in the study if they met any of the following criteria: 1) Coronary angiography (CA) or multi-slice CT coronary angiography (CTCA) suggestive of moderate to severe coronary artery stenosis. 2) Chest tightness, onset of shortness of breath, and poor exercise tolerance after receiving formal drug treatment (with or without stent or bypass graft). 3) Hospitalized more than 2 times within 1 year due to the aforementioned problems. 4) CCS angina grading higher than grade II, and NYHA functional classification of I-III. 5) More than 1 month after acute myocardial infarction (AMI) and more than 2 weeks after PCI surgery. The diagnosis and treatment in all the patients was in accordance with the related domestic and European guidelines developed in 2007

ELIGIBILITY:
Inclusion Criteria:

* coronary angiography or multi-slice spiral ct coronary angiography suggestive of moderate to severe coronary artery stenosis.
* Chest tightness, onset of shortness of breath, and poor exercise tolerance after receiving formal drug treatment with or without stent or bypass graft).
* Hospitalized more than 2 times within 1 year due to the aforementioned problems.
* Canadian Cardiovascular Society angina grading higher than grade II, and New York Heart Association functional classification of I-III.
* More than 1 month after acute myocardial infarction (AMI) and more than 2 weeks after PCI surgery. The diagnosis and treatment in all the patients was in accordance with the related domestic and European guidelines developed in 2007.

Exclusion Criteria:

* Acute myocardial infarction or coronary artery bypass graft within the 4 weeks prior to the study.
* History of heart transplantation.
* History of metal valve replacement surgery.
* Intracardiac thrombus.
* Left ventricular ejection fraction < 30% and unstable hemodynamics.
* Arrhythmia with a rate < 40 bpm or > 120 bpm.
* Skin ulceration or infection in the treatment area.
* Severe obstructive lung disease.

Ages: 35 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Extracorporeal Cardiac Shock Wave Therapy (CSWT) for Treatment of Coronary Artery Disease | 3 years
  Outcome measure included clinical assessment and morphological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Guo Tao, MD, Study Director — Kunming Medical University
Locations (1):
- Cardiovascular Center, Kunming, Yunnan, China

REFERENCES:
- [Derived] Nirala S, Wang Y, Peng YZ, Yang P, Guo T. Cardiac shock wave therapy shows better outcomes in the coronary artery disease patients in a long term. Eur Rev Med Pharmacol Sci. 2016;20(2):330-8. PMID 26875905